CLINICAL TRIAL: NCT05343377
Title: Prospective, Multicenter Clinical Study of Accurate Stratification and Prognostic Value of Circulating Free Methylated EBV DNA in Extranodal NK/T Cell Lymphoma
Brief Title: A Clinical Study of the Value of Circulating Free Methylated EBV DNA in Extranodal NK/T Cell Lymphoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Zhenjiang First People's Hospital (Other); Changzhou First People's Hospital (Unknown); Changzhou Second People's Hospital (Unknown); Wuxi People's Hospital (Other); Second Affiliated Hospital of Soochow University (Other); The First Affiliated Hospital of Nantong University (Unknown); Huaian first people's hospital (Unknown); Yancheng First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB-GL1-AF02
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Extranodal Natural Killer/T-cell Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- circulate free methylated EBV DNA predicts PFS rate in ENKTCL (Experimental)
  Interventions: Diagnostic Test: circulate free methylated EBV DNA

INTERVENTIONS:
Diagnostic Test: circulate free methylated EBV DNA — Accuracy of circulating free methylated EBV DNA in predicting 2-year PFS

SUMMARY:
This study is a prospective, multicenter, open-label, single-arm clinical study. This study plans to enroll 72 newly diagnosed ENKTCL patients. The enrollment was completed in 2 years, and the follow-up was terminated in 4 years. To observe the accuracy of circulating free methylated EBV DNA in predicting 2-year PFS rate, 2-year OS rate, and CR rate in newly diagnosed ENKTCL patients; and to clarify the prognostic stratification ability of PINK-cpgE compared with PINK-E

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed ENKTCL confirmed by pathological tissue, the diagnostic criteria refer to the 2016 WHO diagnostic criteria
* Sign written informed consent and be able to comply with the visits and related procedures specified in the protocol

Exclusion Criteria:

* The investigator believes that the subjects may have other factors that may affect the efficacy or safety evaluation of this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessing the accuracy of circulating free methylated EBV DNA in predicting 2-year PFS in patients with newly diagnosed ENKTCL | 2 years

SECONDARY OUTCOMES:
To assess the accuracy of circulating free methylated EBV DNA in predicting 2-year OS and CR rates in newly diagnosed ENKTCL patients | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, China

IPD SHARING:
Plan to Share IPD: Undecided